CLINICAL TRIAL: NCT07215975
Title: REal-World Application of Luspatercept in Adults With Transfusion-Dependent Beta-Thalassemia in the Middle East (RELATE): A Non-interventional Retrospective and Prospective Observational Study
Brief Title: A Real-World Study to Evaluate Luspatercept in Adults With Transfusion-Dependent Beta-Thalassemia in the Middle East
Status: Not yet recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1107
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: β-thalassemia
Keywords: Transfusion-dependent β-thalassemia
MeSH Terms: interventions — luspatercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Participants receiving luspatercept treatment
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — According to the product label

SUMMARY:
The purpose of this study is to evaluate luspatercept treatment in adults with transfusion-dependent beta-Thalassemia in the Middle East

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants of any race aged at least 18 years at time of initiation of luspatercept treatment
* Participants with documented diagnosis of transfusion-dependent β-thalassemia (TDT).
* Participants who have been initiated on treatment with luspatercept as per the product's Summary of Product Characteristics (SmPC) no longer than 12 months prior to informed consent signature, and for whom therapy is ongoing.
* Participants for whom the decision to prescribe luspatercept treatment is clearly separated from the physician's decision to include the participant in the current study.
* Participants who have provided signed informed consent for participating in the study and for collecting and analyzing medical data pertinent to the objectives of this study

Exclusion Criteria:

* Participants that meet any of the contraindications to the administration of luspatercept as outlined in the latest version of the locally approved SmPC.
* Participants who are currently receiving or are planned to receive treatment with any investigational drug/device/intervention or who have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) prior to luspatercept therapy initiation.
* Participants who are currently pregnant, breastfeeding, or planning a pregnancy during the study observation period.
* Participants who have not provided signed informed consent for participating in the study and for collecting and analysing medical data pertinent to the objectives of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients with transfusion-dependent β-thalassemia (TDT) in the Middle East region who have initiated luspatercept treatment
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-25 (Estimated); Primary Completion 2030-02-28 (Estimated); Study Completion 2031-04-17 (Estimated)

PRIMARY OUTCOMES:
Change in transfusion burden | Baseline and up to week 144
Change in mean pre-transfusion hemoglobin level | Baseline and up to week 144

SECONDARY OUTCOMES:
Change in transfusion-related visits | Baseline and up to week 144
Proportion of participants achieving ≥33% reduction in red blood cell (RBC) transfusion burden (number of RBC units transfused) plus a reduction of ≥2 units | Baseline and up to week 144
Proportion of participants achieving ≥50% reduction in red blood cell transfusion burden plus a reduction of ≥2 units | Baseline and up to week 144
Time from first luspatercept dosing date to the first erythroid response | Baseline and up to week 144
Time from the date the erythroid response is first observed until the last day of response | Baseline and up to week 144
Participant pretransfusion hemoglobin level | Baseline and up to week 144
Participant baseline transfusion burden | Baseline
Proportion of participants without red blood cell transfusion during any consecutive 12-week or 24-week treatment period | Baseline and up to week 144
Time from first luspatercept dosing date to first onset of red blood cell-transfusion independence ≥12 weeks and ≥24 weeks | Baseline and up to week 144
Time from the date a 12-week and 24-week red blood cell-transfusion independence is first observed until the date the participant has a subsequently documented red blood cell transfusion | Baseline and up to week 144
Change in mean serum ferritin (SF) level | Baseline and up to week 144
Change in proportion of participants with mean serum ferritin <1,000, 1000-2500, and >2,500 μg/L | Baseline and up to week 144
Types (drug formulation - mono and combination therapy) of iron chelation therapy received | Baseline and up to week 144
Change in mean daily dose of iron chelation therapy from baseline | Baseline and up to week 144
Number of medical encounters (inpatient hospitalizations, emergency department attendances, hospital outpatient visits, visits at office-based physicians) | Baseline and up to week 144
Inpatient length of stay | Baseline and up to week 144
Proportion of participants remaining on luspatercept treatment | Up to week 144
Length of time from initiation to discontinuation of luspatercept treatment | Up to week 144
Frequencies of reasons for discontinuation of luspatercept treatment | Up to week 144
Participant sociodemographics | Baseline
  Sociodemographics of participants such as age, sex, ethnicity, country of treatment, height, weight, and body mass index
Participant disease characteristics | Baseline
  Disease characteristics of participants, describing age of diagnosis of β-thalassemia, genotype (β0/β0, non-β0/β0), splenectomy status (yes/no), pretransfusion hemoglobin level (mean of all documented), transfusion burden (total number of red blood cell units transfused).
Participant comorbidities | Baseline
  Disease- and non-disease-related comorbid conditions
Concomitant treatment(s) received | Baseline
  Disease-related best supportive care (BSC) and treatments for other comorbidities.
Number of luspatercept doses administered | Up to week 144
Number of luspatercept dose modifications | Up to week 144
Frequencies of reasons for luspatercept dose modifications | Up to week 144

CONTACTS AND LOCATIONS:
Overall Officials: Bristol Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Prince Muhammad bin Nasser Hospital, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts